CLINICAL TRIAL: NCT06494306
Title: Characterization of Olfactory Perception in Post-Traumatic Stress Disorder
Acronym: TRAUMODO
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0189
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post traumatic stress disorder; Olfactory perception; Olfaction; Odor
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anosmia | interventions — Surveys and Questionnaires; Odorants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with PTSD: They are outpatients receiving psychological and medical treatment in the clinical department connected to the inclusion site
  Interventions: Behavioral: European Test of Olfactory Capabilities (ETOC); Behavioral: Standardized Hedonicity Test; Behavioral: Questionnaires; Behavioral: Odor / trauma association questionnaire
- Control group: Data from subjects without PTSD included in a previous study
  Interventions: Behavioral: European Test of Olfactory Capabilities (ETOC); Behavioral: Standardized Hedonicity Test

INTERVENTIONS:
Behavioral: European Test of Olfactory Capabilities (ETOC) — Investigators will collect the ETOC score in patient of both arms
Behavioral: Standardized Hedonicity Test — To smell 20 odorant solutions and for each odor and evaluate it along five dimensions: familiarity, hedonicity, edibility, desire to smell again, perceived intensity). Each dimension is assessed with a Likert scale (from 1 (not at all) to 9 (extremely))
Behavioral: Questionnaires — Patients with PTSD will have the following questionnaires : PTSD Checklist for Diagnostic and Statistical Manual (DSM)-V (PCL-5), Peri-trauma Dissociation Experience Questionnaire (PDEQ), Patient Health Questionnaire-9 (PHQ9), Snaith-Hamilton Pleasure Scale (SHAPS), Childhood Trauma Questionnaire (CTQ) and Apathy Evaluation Scale (AES)
  Groups: Patients with PTSD
Behavioral: Odor / trauma association questionnaire — Patients with PTSD will have Odor / trauma association questionnaire
  Groups: Patients with PTSD

SUMMARY:
The core symptoms of post-traumatic stress disorder (PTSD) include flash backs, intrusive pictures and thoughts related to the traumatic event, hyperalertness, avoidance of traumatic relevant environmental triggers and emotional dysregulation. Some studies suggest that PTSD is also associated with impaired olfactory perception, which seems quite intuitive regarding the close anatomical-functional connections between olfactory and emotional circuits. Furthermore, some studies reported that olfactory stimuli can trigger flashbacks in subjects with PTSD. However, up to know available data is scarce and heterogeneous concerning that topic. The goal of the study is to determine the olfactory phenotype of subjects with PTSD. More precisely, this project aims at filling the above mentioned gap by systematically assessing the olfactory perception of subjects with PTSD along five dimensions: olfactory identity, hedonic value, familiarity, desirability and edibility. As a secondary goal, the relative weight of olfaction compared to the other senses in the relived memories of subjects with PTSD will be assessed.

The investigators here hypothesize a global impairment in olfactory processing (intensity, hedonicity, familiarity and edibility judgments) in PTSD subjects, compared with healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 50
* Subjects with PTSD

Exclusion Criteria:

* Patients with a neurological history such as stroke, head trauma (e.g. exposure to explosions, sports injury…), neurodegenerative disease…
* Any psychiatric condition except PTSD and major depressive disorder
* Current or recent use of psychotropic drugs that may affect olfactory function.
* Any current or remitted addictive disorder.
* Pregnancy and breast-feeding women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients aged 18 to 50 suffering from PTSD
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-08-26 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Standardized Hedonicity Test score | at inclusion
  Results obtained in patients will be compared to those obtained in control group

SECONDARY OUTCOMES:
Effects of potential moderators on odor judgement | at inclusion
  Analysis of covariance (ANCOVA) to determine the effect of different moderators (age, gender, type of trauma, time elapsed since trauma, type of treatment received, symptom intensity) on olfactory perception
Evaluation of sensory impressions of memories evoked by certain odors. | at inclusion
  Sensory impressions: Nature and frequency of sensory descriptions associated with odor-evoked memories
Evaluation of emotional valence of memories evoked by certain odors. | at inclusion
  Language analysis: Use of Natural Language Processing (NLP) techniques to assess the emotional valence of odor-evoked memories and recurrent themes in oral responses concerning evoked memories. Analysis of the association of trauma-related odors with the 5 senses

CONTACTS AND LOCATIONS:
Overall Officials: VIGNAUD Philippe, MD, PhD, Principal Investigator — Auvergne-Rhône-Alpes Regional Center for Psychotrauma
Locations (1):
- Auvergne-Rhône-Alpes Regional Center for Psychotrauma, Lyon, France

IPD SHARING:
Plan to Share IPD: No